CLINICAL TRIAL: NCT04177589
Title: Incidence of Delirium and Some Related Factors in Elderly Patients Hospitalized in Geriatrics Department, Gia Dinh Hospital.
Brief Title: Incidence of Delirium in Inpatient Elderly Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, Dinh Pham Thi Thuy Van, MD, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: NTL
Record Dates: First submitted 2019-11-24; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Incidence of Delirium in Inpatient Elderly Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Incidence of Delirium in Inpatient Elderly Patients — Study design: prospective cohort study.

SUMMARY:
Study: prospective cohort study Register for research topic on ClinicalTrails.gov. Convenience sampling, all patients aged 60 and older entered the geriatric department of Gia Dinh People's Hospital in Ho Chi Minh City from December 2020 to May 2021.

Direct interview with the patient. Minimum time 10-15 minutes for each interview.

Evaluation at the time of admission (within the first 24 hours of admission): demographic characteristics, diagnosis at Geriatric ward, frailty, activities of daily living.

Assessment during hospital stay: identifying delirum using the CAM tool. Assessment at the time of discharge: diagnosis at discharge and the drugs used during inpatient treatment in the department.

Research objectives:

1. Determine the incidence of delirium in elderly patients in general geriatric department.
2. Investigate some of the important related factors that are common for delirium in elderly patients in general geriatric department.
3. Determine the relationship between delirium and clinical outcomes in elderly patients in general geriatric department.

DETAILED DESCRIPTION:
Study design: prospective cohort study. Time: From December 2020 to May 2021. Place: Department of Geriatrics, Gia Dinh People's Hospital, Ho Chi Minh City. Sample population: All patients aged 60 and older entered the Geriatric Department of Gia Dinh People's Hospital in Ho Chi Minh City from December 2020 to May 2021.

Sampling technique: Convenience sampling Admission criteria: All patients ≥ 60 years of age agree to participate in the study.

Exclusion criteria: Disturbance or other cognitive disorders at the time of assessment at admission, hospital stay not exceeding 48 hours

Data collection:

Data collection process:

Direct interview with the patient. Minimum time 10-15 minutes for each interview (excluding time to explain purpose, method of conducting research, time for collecting information on demographic characteristics and medical conditions).

Person doing interview: geriatric resident doctors including Dinh Pham Thi Thuy Van, Huynh Khoi Nguyen, Tran Tan Dat The interviewers will explain the research objectives and only started conducting the interview when the patient or his relative (authorized) agreed to participate in the study.

Conduct interviews:

*Evaluation at the time of admission (within the first 24 hours of admission): Patients entering the geriatric ward who agree to participate in the study will be assessed by the doctor for cognitive status, clinical characteristics and a diagnostic flow chart for Delirium

Record details about:

* Demographic characteristics: gender, age, address, occupation, family status and marital status.
* Diagnosis at the time of admission, co-morbidities (pulmonary disease, hypertension, type 2 diabetes, chronic kidney disease, osteoporosis, osteoarthritis, constipation, liver and gastrointestinal diseases, cardiovascular disease, arrhythmia, endocrine and metabolic disorders, neurological diseases, urological diseases, hematological pathologies and other diseases). Amount and type of medication being taken at home up to the time of admission. Routine tests.
* Frailty status, functional activities according to ADLs and IADLs scale, initial cognitive status according to MMSE, vision and hearing.

  * Evaluation during the hospital stay:

When a patient is suspected of delirium, we evaluate it using the CAM tool to identify. After that, the patient was recorded the following characteristics: the time of onset, the clinical form (increased activity, decreased activity or mixed), current medical conditions and medications.

Record falls, transfer to other wards (if any).

*Evaluation at the time of discharge: At the time of discharge, we will record the time of hospitalization, the reason for discharge (improved condition or relative request due to serious illness) or the place of hospital transfer or in-hospital death (if any).

Record diagnosis on discharge and drugs used during inpatient treatment at the department

Data collection tools: A sheet of prepared data and medical records.

Bias control:

* Information discrepancy

  * Clearly define the subjects of study.
  * Choose a sample according to admission and exclusion criteria
* Selection errors

  * The person doing the interview is the person who wrote the data collection sheet, so it will limit the errors in the interview process.
  * The variables are clearly defined and measurable.
  * Collect information in a unified form.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 60 years of age agree to participate in the study.

Exclusion Criteria:

* Disturbance or other cognitive disorders at the time of assessment at admission, hospital stay not exceeding 48 hours

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients aged 60 and older entered the Geriatric Department of Gia Dinh People's Hospital in Ho Chi Minh City from December 2020 to May 2021.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-12-15 (Estimated); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-08-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Delirium in Inpatient Elderly Patients | from December 2020 to May 2021
  Incidence of Delirium in elderly patients entered the Geriatric Department of Gia Dinh People's Hospital in Ho Chi Minh City

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatrics, Gia Dinh People's Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No